CLINICAL TRIAL: NCT00190892
Title: Olanzapine Plus Carbamazepine Versus Carbamazepine Alone in the Treatment of Manic or Mixed Episodes Associated With Bipolar I Disorder
Brief Title: Olanzapine Plus Carbamazepine in the Treatment of Bipolar I Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7031; F1D-MC-HGKR
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine; Carbamazepine

INTERVENTIONS:
Drug: olanzapine
Drug: carbamazepine

SUMMARY:
This trial will assess any efficacious benefit and any safety issues associated with the concomitant use of olanzapine and carbamazepine for the treatment of patients with bipolar I disorder, manic or mixed episodes

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of bipolar disorder and currently meet DSM-IV-TR criteria for a manic or mixed episode
2. Female patients must test negative on a serum pregnancy test at the time of enrollment and agree to use medically accepted contraception throughout the study.
3. Have YMRS score > or = 20 at both the screening (Visit 1) and randomization (Visit 2) visits.

Exclusion Criteria:

1. Have participated (been randomized) in a clinical trial of another investigational drug (including olanzapine or carbamazepine) within 30 days prior to Visit 1
2. Have a history of agranulocytosis (absolute neutrophil count< 500/uL) during the patient's lifetime
3. Have acute, serious or unstable medical conditions, including (but not limited to) inadequately controlled diabetes (HgbA1c>8%); severe hypertriglyceridemia (fasting triglycerides > or = 500 mg/dl;hepatic insufficiency (specifically any degree of jaundice); recent cerebrovascular accidents; uncontrolled seizure disorders; serious acute systemic infection or immunologic disease: unstable cardiovascular disorders (including ischemic heart disease); or renal, gastroenterologic, respiratory, endocrinologic, neurologic, or hematologic diseases (specifically current absolute neutrophil count , <1500/uL)
4. Have a substance dependence (except nicotine or caffeine), based on DSM-IV-TR criteria, within the 30 days prior to study entry.
5. Require concomitant treatment with any other medication with primarily central nervous system (CNS) activity, other than those allowed in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-09; Study Completion 2006-06

PRIMARY OUTCOMES:
To assess the superiority of olanzapine plus carbamazepine versus placebo plus carbamazepine in improving overall manic symptomatology in patients with mania associated with bipolar I disorder.
Improvement is measured by a reduction in the total score of the Young Mania Rating Scale (YMRS) from baseline to endpoint during the 6-week, double-blind treatment phase.

SECONDARY OUTCOMES:
To compare the efficacy and safety of up to 6 weeks of double-blind, concomitant use of olanzapine plus carbamazepine to the concomitant use of placebo plus carbamazepine
Using the following assessments:
rate of response and time to response over 6 weeks of the double-blind treatment phase, with response defined as a reduction of 50% or more in the YMRS total score from baseline to endpoint.
rate of remission and time to remission of mania over 6 weeks of the double-blind treatment phase, with remission defined as a score less than or equal to 12 on the YMRS total score at endpoint
reductions from baseline to the endpoint of the 6-week, double-blind treatment phase on the Montgomery-Asberg Depression Rating Scale (MADRS) total score
reductions from baseline to the endpoint of the 6-week, double-blind treatment phase on the Clinical Global Impressions-Bipolar Version Severity of Illness Scale (CGI-BP)score
rate of switch to depression and time to switch to depression, with switch to depression defined as a baseline MADRS total score less than or equal to 12 followed by
either a post baseline MADRS total score greater than or equal to 16 over the 6 weeks of the double-blind treatment phase OR, hospitalization due to deterioration in clinical
symptoms of depression
longitudinal effects from baseline across visits of the double-blind treatment phase by comparing changes in YMRS total scores
changes in vital signs and weight, laboratory analytes, and electrocardiograms (ECGs), and the incidence and severity of TEAEs and extrapyramidal symptoms (EPS)
using the Barnes Akathisia Scale, Simpson-Angus Scale and the AIMS.
the effect of carbamazepine on the plasma concentration of olanzapine via comparison to historic oral steady-state olanzapine concentrations
the effect of olanzapine on the plasma concentrations of carbamazepine via a descriptive comparison of the two treatment groups
Additional secondary objectives are to assess the maintenance of treatment effect and safety of up to 20 weeks of open-label olanzapine-plus-carbamazepine treatment
using the following measures:
YMRS total score change from the baseline (Visit 7) to the endpoint of the open-label treatment phase.
rate of relapse to mania during the open-label treatment phase. Relapse to mania (patients who relapse to a bipolar I mania or mixed episode) is defined by the following:
patient reaches remission of mania (as defined by a YMRS score less than or equal to 12) by the endpoint of the double-blind treatment phase
patient obtains a YMRS score greater than or equal to 15 at any time during the open label treatment phase AND/OR becomes hospitalized due to deterioration in clinical symptoms of mania
rate of switch to depression during open-label treatment phase, with switch to depression defined as a baseline MADRS total score less than or equal to 12 followed by
either a postbaseline MADRS total score greater than or equal to 16 over the 20 weeks of the open-label treatment phase hospitalization due to deterioration in clinical symptoms of depression
changes in vital signs and weight, laboratory analytes, and ECGs, and the incidence and severity of TEAEs and EPS using the Barnes Akathisia Scale, Simpson-Angus Scale, and the Abnormal Involuntary Movement Scale (AIMS)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Everton Park, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Epping, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Frankston, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Malvern, Victoria
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Corfu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kavala
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tripoli
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Gyula
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Székesfehérvár
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Saint Petersburg

REFERENCES:
- [Derived] Tohen M, Bowden CL, Smulevich AB, Bergstrom R, Quinlan T, Osuntokun O, Wang WV, Oliff HS, Martenyi F, Kryzhanovskaya LA, Greil W. Olanzapine plus carbamazepine v. carbamazepine alone in treating manic episodes. Br J Psychiatry. 2008 Feb;192(2):135-43. doi: 10.1192/bjp.bp.107.041301. PMID 18245032